CLINICAL TRIAL: NCT00261586
Title: Effect of Analgesics on the Irreversible Inactivation of Cyclooxygenase-1 Activity by Low Dose Aspirin and Endoscopic Evaluation of the Gastric Mucosal Effect
Brief Title: A Safety Trial to Compare Different Analgesics in Combination With Low Dose Aspirin to Study Their Bleeding Properties and Their Effects on the Stomach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR002500
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Analgesics
Keywords: aspirin; analgesics; cyclooxygenase activity; non-steroidal antiinflammatory drugs
MeSH Terms: interventions — Aspirin; Acetaminophen; Ibuprofen; Naproxen; Celecoxib; rofecoxib

INTERVENTIONS:
Drug: aspirin, acetaminophen, ibuprofen, naproxen, celecoxib, rofecoxib

SUMMARY:
The purpose of this study is to compare several analgesics given in approved daily doses in combination with a daily cardioprotective dose of aspirin (81 mg), to study their bleeding properties and their effects on the stomach in healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this randomized, multiple-dose, single-blind, parallel-group study is to examine in healthy volunteers the effects of analgesics given in approved daily doses in addition to daily cardio-protective doses of aspirin (81 mg) on the stomach. All subjects are examined endoscopically before receiving study medication, and at the end of treatment on Day 9. Each subject takes 81 mg of aspirin daily plus one of the following treatments to be taken daily on Days 1 through 8: four doses of acetaminophen 1000 mg, three doses of ibuprofen 400 mg, two doses of naproxen sodium (440 mg in the morning and 220 mg in the evening), four doses of aspirin 650 mg, two doses of celecoxib 200 mg, one dose of rofecoxib 25 mg, or no additional study medication. On Day 9, one dose of aspirin 81 mg and only one dose of the assigned treatment drug are taken prior to having an endoscopy. The primary endpoints of the study are the effects of the analgesics on the inhibition of COX-1 activity by aspirin, and any injury to the stomach mucosa, as determined by direct endoscopic observation. Safety assessments consist of routine monitoring for adverse events, as well as endoscopic examination of gastric mucosa for erosions and ulcerations occurring during the treatment phase. The study hypothesis is that the effects of acetaminophen on the stomach do not differ from the effects of ibuprofen, naproxen, aspirin, celecoxib, or rofecoxib. 81 mg aspirin and 1of 7 treatments for 8 days: acetaminophen 1000mg 4xday, ibuprofen 400mg 3xday, naproxen 440mg morning and 220mg evening, no additional study medication, aspirin 650mg 4xday, celecoxib 200mg 2xday,rofecoxib 25mg 1xday. On Day 9, 1 dose aspirin & 1 dose study drug before endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* In general good health with normal hemostatic (blood coagulation) parameters
* able to swallow study medication
* non-smoker
* negative for H. pylori infection
* if female, must not be pregnant or breast feeding

Exclusion Criteria:

* Have taken anti-inflammatory drugs within one week of study entry, any analgesic within 24 hours before baseline endoscopy, or systemic steroids within 6 weeks of study entry
* unable to tolerate oral drugs or have had gastrointestinal disease or prior gastrointestinal surgery that could interfere with the study medication
* unable to understand or follow instructions
* have a medical condition or clinically significant abnormal laboratory results that may be relevant to participation in the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Percent arachidonic acid-induced platelet aggregation; Lanza Mucosal Injury Score of the stomach

SECONDARY OUTCOMES:
Serum thromboxane B2; plasma PGE2; shear-induced platlet aggregation; cyclooxygenase activity in stomach mucosal biopsies as assessed by PGE2 content

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: A Safety Trial to Compare Different Analgesics in Combination with Low Dose Aspirin to Study Their Bleeding Properties and Their Effects on the Stomach — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=906&filename=CR002500_CSR.pdf